CLINICAL TRIAL: NCT07289165
Title: Comparison of Pharmacokinetic Responses to Three Ketone Esters
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NeuroEnergy Ventures, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: NE-01-2025
Record Dates: First submitted 2025-12-03; First posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Healthy Volunteer

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 12.5mg Ketone Tri Ester (Active Comparator): Dietary Supplement containing Tri-betahydroxybutyrin
  Interventions: Dietary Supplement: Dietary Supplement containing Tri-betahydroxybutyrin
- 12.5mg Ketone Mono Ester (Active Comparator): Dietary Supplement containing a ketone mono Ester
  Interventions: Dietary Supplement: Dietary Supplement containing a ketone mono Ester
- 12.5mg Ketone Salt (Active Comparator): Dietary supplement containing a ketone salt
  Interventions: Dietary Supplement: Dietary supplement containing a ketone salt

INTERVENTIONS:
Dietary Supplement: Dietary Supplement containing Tri-betahydroxybutyrin — Ketone Tri Ester
  Arms: 12.5mg Ketone Tri Ester
Dietary Supplement: Dietary Supplement containing a ketone mono Ester — Ketone Mono Ester
  Arms: 12.5mg Ketone Mono Ester
Dietary Supplement: Dietary supplement containing a ketone salt — Dietary Supplement from a ketone salt
  Arms: 12.5mg Ketone Salt

SUMMARY:
The purpose of this study is to examine how the body absorbs, digests, and metabolizes three different investigational ketone dietary supplements (ketone monoester, ketone tri-ester, ketone salt) and to assess gastrointestinal tolerance or other adverse effects. This study is considered investigational because data are being collected on the differences over time between three active study products. Consumption of these study products are not intended to diagnose, treat, cure, or prevent any disease.

DETAILED DESCRIPTION:
* This study is a randomized, double-blind, crossover trial of N=18 apparently healthy men and women between 30 and 70 years old to be recruited at a single investigational center.
* Participants will attend 7 study visits. During Visit 1 participants will be screened for eligibility [i.e., medical history, routine blood work, background baseline diet]. During visits 2, 4, and 6 participants will undergo consumption of a study product (either ketone monester, ketone triester, or ketone salt) and serial blood draws for serum beta-hydroxybutyrate (BHB) will be used to assess the pharmacokinetic (PK) response over an 8-hour period with an additional 24-hour post-ingestion blood draw (to occur on visits 3, 5 and 7). In addition, participants will rate their overall GI tolerance, alertness, and focus via visual analog scales (VAS). During visits 3, 5 and 7 (which will be 24 hours after visits 2, 4, and 6, respectively) participants will undergo a single blood draw for BHB at the 24-hour post ingestion time point and rate their overall GI tolerance via VAS.
* Comprehensive side effect profile/ adverse event monitoring will take place throughout the study duration. The study will be conducted following ICH-GCP guidelines to ensure subject safety and scientific integrity of the data.

ELIGIBILITY:
Inclusion Criteria:

* • Provide voluntary signed and dated informed consent.

  * Be in good health as determined by medical history and routine blood chemistries.
  * Age between 30 and 70 yr (inclusive).
  * Body Mass Index of 25-34.9 (inclusive).
  * Body weight of at least 120 pounds.
  * Normotensive (seated, resting systolic blood pressure <140 mm Hg and diastolic blood pressure < 90 mm Hg. If the first measurement is slightly elevated above these limits, the subject will be given a brief (5 minute) rest period, and two more measurements will be taken. The average of all three measurements will be used to determine eligibility.
  * Normal seated, resting heart rate (<90 per minute).
  * Willing to duplicate and record their previous 24-hour diet, refrain from caffeine, alcohol and exercise for 24 hours prior to each visit, and fast for 10 hours prior to each visit.
  * Subject agrees to maintain existing dietary and physical activity patterns throughout the study period.
  * Subject is willing and able to comply with the study protocol.

Exclusion Criteria:

* Individuals using any kind of GLP-1 medications.

  * Individuals who are determined to have liver, renal, cardiovascular, neurological, or other metabolic disease.
  * History or presence of diabetes, prediabetes or endocrine disorder.
  * Use of any dietary supplements or medications which may confound the study or its endpoints (e.g., fish oil, choline donors, gingko biloba, phosphatidylserine, huperzine A, etc.).
  * Alcohol consumption (more than 2 standard alcoholic drinks per day or more than 10 drinks per week) or drug abuse or dependence within the past 6 months.
  * Current nicotine use > 100 mg/day.
  * History of hyperparathyroidism or an untreated thyroid condition.
  * History of malignancy in the previous 5 years, except for non-melanoma skin cancer (basal cell cancer or squamous cell cancer of the skin).
  * History of chronic psychiatric conditions (e.g., bipolar, schizophrenia, PTSD, depression, etc.).
  * History of brain disorders [e.g., stroke, MS, Parkinson's, history of TBI or epilepsy, migraine (>1 migraine per month), etc.].
  * Prior gastrointestinal bypass surgery (Lapband), etc.
  * Other known gastrointestinal or metabolic conditions that might impact nutrient absorption or metabolism, e.g., short bowel syndrome, Inflammatory bowel syndrome (IBS), Inflammatory bowel disease (IBD; e.g., Crohn's, ulcerative colitis), diarrheal illnesses, history of colon resection, gastro paresis, Inborn-Errors-of-Metabolism (such as PKU).
  * Chronic inflammatory condition (e.g., rheumatoid arthritis, Lupus, HIV/AIDS, etc.).
  * Previous medical diagnosis of asthma, gout, or fibromyalgia.
  * Currently following a low-carbohydrate, keto type diet, or practicing an intermittent fasting lifestyle (>14 hours of fasting).
  * Subjects that have donated blood or plasma within the previous week.
  * Pregnant women, women trying to become pregnant, women less than 120 days postpartum or nursing women. Women who participate in this study must agree to the use of contraception for the duration of the study and any woman that is sexually active will have to take pregnancy test prior to enrolling with a negative result. Women of childbearing age (any woman prior to menopause) regardless of their use of contraception will be provided a urine pregnancy test kit at their screening visit and take the test in private using the female lavatory after signing an informed consent.
  * Known sensitivity to any ingredient in the test formulations as listed in the product label.
  * Currently participating in another research study with an investigational product or have been in another research study in the past 30 days.
  * Clinically significant abnormal laboratory results at screening.
  * Any other conditions that, in the opinion of the medical staff, could confound the primary endpoints or place the subject at increased risk of harm if they were to participate.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2025-07-15 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Serum BHB concentration maximum (Cmax) | blood draws will be performed before (0 min) and 15-, 30-, 45-, 60-, 90-, 120-, 150-, 180-, 240-, 300-, 360-, and 480 min post ingestion of the study product
time to maximum concentration (Tmax) | blood draws will be performed before (0 min) and 15-, 30-, 45-, 60-, 90-, 120-, 150-, 180-, 240-, 300-, 360-, and 480 min post ingestion of the study product
area under the curve (AUC), | blood draws will be performed before (0 min) and 15-, 30-, 45-, 60-, 90-, 120-, 150-, 180-, 240-, 300-, 360-, and 480 min post ingestion of the study product
elimination half-life (T1/2), | blood draws will be performed before (0 min) and 15-, 30-, 45-, 60-, 90-, 120-, 150-, 180-, 240-, 300-, 360-, and 480 min post ingestion of the study product
oral clearance | blood draws will be performed before (0 min) and 15-, 30-, 45-, 60-, 90-, 120-, 150-, 180-, 240-, 300-, 360-, and 480 min post ingestion of the study product
volume of distribution | blood draws will be performed before (0 min) and 15-, 30-, 45-, 60-, 90-, 120-, 150-, 180-, 240-, 300-, 360-, and 480 min post ingestion of the study product

SECONDARY OUTCOMES:
Visual Analogue Scale for GI tolerance | assessed at 15-, 30-, 45-, 60-, 90-, 120-, 150-, 180-, 240-, 300-, 360-, and 480 min post ingestion of the study product
Safety (vital signs) and Adverse Events | assessed at 15-, 30-, 45-, 60-, 90-, 120-, 150-, 180-, 240-, 300-, 360-, and 480 min post ingestion of the study product

CONTACTS AND LOCATIONS:
Overall Officials: Tim Ziegenfuss, PhD, Principal Investigator — CAHS
Locations (1):
- CAHS, Canfield, Ohio, United States

IPD SHARING:
Plan to Share IPD: No